CLINICAL TRIAL: NCT01781988
Title: The Clinical Study of Personalized Therapy for Non-small Cell Lung Cancer Based on ERCC1/RRM1/TS Expression
Brief Title: Personalized Therapy in Non-small Cell Lung Cancer
Acronym: PTINCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Heyuwen, Yuwen He, MD, Guangzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZMC12521; PT12521 (Other: The First Affiliated Hospital of Guangzhou Medical University)
Record Dates: First submitted 2013-01-24; First posted 2013-02-01 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Lung Cancer; Carboplatin Adverse Reaction
Keywords: lung cancer; gemcitabine; carboplatin; pemetrexed
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A.individual therapy (Experimental): Carboplatin was administrated at an area under the plasma concentration time curve (AUC) of 5 on day 1 every 21 days, while gemcitabine was administrated at a dose of 1250 mg/m2 on day 1 and 8 and pemetrexed was administrated at a dose of 500 mg/m2 on day 1.
  Interventions: Drug: carboplatin, gemcitabine , pametrexed
- B. non-individualized therapy (Experimental): Carboplatin was administrated at an area under the plasma concentration time curve (AUC) of 5 on day 1 every 21 days, while gemcitabine was administrated at a dose of 1250 mg/m2 on day 1 and 8 and pemetrexed was administrated at a dose of 500 mg/m2 on day 1.
  Interventions: Drug: carboplatin, gemcitabine , pametrexed

INTERVENTIONS:
Drug: carboplatin, gemcitabine , pametrexed — A.individual therapy :enrolled patients with ERCC1 negative tumors who received carboplatin and a third-generation agent (gemcitabine or pametrexed) based on RRM1 or TS expression. If RRM1 protein was negatively expressed in the tumor tissues, gemcitabine was used, whereas pemetrexed was used if RRM1 was positively expressed and TS was negatively expressed.
  B.non-individualized therapy :enrolled patients who received carboplatin and a third-generation agent but were not based on ERCC1, RRM1, or TS expression.

SUMMARY:
Excision repair cross complementing 1 (ERCC1) ribonucleotide reductase M1 (RRM1) and thymidylate synthase(TS) are molecular determinants that predict sensitivity or resistance to platinum agents 、 gemcitabine and pemetrexed respectively.

Tailored therapy using these molecular determinants suggested patient benefit in a previously reported phase 2 trial. Here, we designed a study for an individual patient analysis of prospectively accrued patients who were treated with the "personalized therapy" approach versus other standard approaches.

DETAILED DESCRIPTION:
Patients who had nonsmall- cell lung cancer (NSCLC) performance status of 0/1 were accrued to 2 phase 2 clinical trials Trial A (carboplatin and chemotherapy individuation based on sensitivity marker ), Trial B (carboplatin non-individuation or chemotherapy non-individuation ).

Patients who were treated on Trials B were analyzed as the "standard therapy" group. Patients accrued to Trial A were called the "personalized therapy" group. disease free survival (DFS) was estimated using the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-small cell lung cancer
2. age from 18 years to 75 years
3. ECOG Performance Status no more than 2
4. at least one appraisable lung focus of diameter≥ 10 mm by lung CT
5. Haemoglobin ≥10.0 g/dl, Absolute neutrophil count ≥(ANC) 1.5 x 109/L, platelets ≥100 x 109/L
6. Total bilirubin ≤1.5 x upper limit of normal (ULN)
7. ALT and AST < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases
8. Creatinine clearance ≥60ml/min (calculated according to Cockcroft-gault formula)
9. Informed consent should be obtained before treatment.

Exclusion Criteria:

1. Mixed non-adenocarcinoma cell lung cancer histology
2. Previous treatment for Systemic chemotherapy or local radiotherapy
3. Be allergic to chemotherapy drugs
4. second active primary malignancy or serious concomitant medical disease
5. difficulties with adequate follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The disease-free survival | Followed up these patients for disease-free survival for 4 years
  The disease-free survival was measured from the day of tumor resection until tumor recurrence (progression) or death as the end point

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, Proressor, Study Chair — The first affiliated hospital of Guangzhou MC
Locations (1):
- The first affiliated hospital of Guangzhou MC, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] He YW, Zhao ML, Yang XY, Zeng J, Deng QH, He JX. Prognostic value of ERCC1, RRM1, and TS proteins in patients with resected non-small cell lung cancer. Cancer Chemother Pharmacol. 2015 Apr;75(4):861-7. doi: 10.1007/s00280-015-2714-y. Epub 2015 Mar 3. PMID 25732635